CLINICAL TRIAL: NCT04950543
Title: Effects of an Online Meditation Course on Quality of Life and Positive Emotions - a Prospective Observational Study (EXPAN Study)
Brief Title: Effects of an Online Meditation Course on Quality of Life
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Andreas Michalsen, Principal Investigator, Charite University, Berlin, Germany
Other Study IDs: EXPAN
Record Dates: First submitted 2021-06-10; First posted 2021-07-06 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Quality of Life
Keywords: Meditation
MeSH Terms: interventions — Meditation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Meditation
  Interventions: Behavioral: Meditation

INTERVENTIONS:
Behavioral: Meditation — An online survey will be offered to participants who have enrolled in a 21-day meditation online course. The survey will be conducted using mobile website technology before and after the online course and additionally after 3 and 6 months.

SUMMARY:
Many interventions in the field of meditation are becoming increasingly popular and have gained worldwide acceptance over the past years, both in terms of health, but also psychological aspects. On the other hand, controversial and sometimes hypercritical positions are on the rise, questioning the positive effects of meditation on health due to the limited availability of high-quality scientific data. With regard to a large number of meditation interventions, the systematic exploration of procedures that have not yet been scientifically evaluated - also in online settings - is a meaningful contribution to meditation research.

ELIGIBILITY:
Inclusion criteria:

* Age: 18 years or older
* All persons registering for the online course
* Internet access
* Sufficient language skills, as well as cognitive and physical abilities, to participate in an online survey lasting approximately 30 minutes
* Active consent to the online consent form

Exclusion criteria

- Failure to provide informed consent to participate in the study

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: - All persons registering for the online course
Sampling Method: Non-Probability Sample
Enrollment: 374 (Actual)
Dates: Start 2021-07-05 (Actual); Primary Completion 2021-10-17 (Actual); Study Completion 2021-10-17 (Actual)

PRIMARY OUTCOMES:
Quality of life, PROMIS-29 Profile v2.1 | Change from Baseline Quality of life at 1 months
  The scale ranges from 0 to 100, where 0 is the lowest level and 100 is the highest level.

SECONDARY OUTCOMES:
Quality of life, PROMIS-29 Profile v2.1 | Baseline, 3 months and 6 months
  The scale ranges from 0 to 100, where 0 is the lowest level and 100 is the highest level.
Global Health, PROMIS Scale v1.2 | Baseline, 1 month, 3 months and 6 months
  The scale ranges from 0 to 100, where 0 is the lowest level and 100 is the highest level.
Affect regulation, PANAS 10 | Baseline, 1 month, 3 months and 6 months
  The scale ranges from 1 to 5, where 1 is the lowest level and 5 is the highest level.
Stress, PSS 4 | Baseline, 1 month, 3 months and 6 months
  The scale ranges from 0 to 16, where 0 is the lowest level and 16 is the highest level.
Flourishing, FS 8 | Baseline, 1 month, 3 months and 6 months
  The scale ranges from 8 to 56, where 8 is the lowest level and 56 is the highest level.
Resilience, CD-RISC 10 | Baseline, 1 month, 3 months and 6 months
  The scale ranges from 0 to 4, where 0 is the lowest level and 40 is the highest level.
Mysticism, HMS-8 | Baseline, 1 month, 3 months and 6 months
  The scale ranges from 0 to 100, where 0 is the lowest level and 100 is the highest level.
Self-efficacy, ASKU | Baseline, 1 month, 3 months and 6 months
  The scale ranges from 1 to 5, where 1 is the lowest level and 5 is the highest level.
Awe and Gratitude, GrAw-7 | Baseline, 1 month, 3 months and 6 months
  The scale ranges from 0 to 100, where 0 is the lowest level and 100 is the highest level.
Spirituality, ASP | Baseline, 1 month, 3 months and 6 months
  The scale ranges from 0 to 100, where 0 is the lowest level and 100 is the highest level.
Sedentary behavior | Baseline, 1 month, 3 months and 6 months
  Duration in minutes
Sporting activity | Baseline, 1 month, 3 months and 6 months
  Duration in minutes
Relaxation behavior | Baseline, 1 month, 3 months and 6 months
  Duration in minutes
Alcohol consumption | Baseline, 1 month, 3 months and 6 months
  Assessed retrospectively (last 1 month) with self-designed question
Cigarettes | Baseline, 1 month, 3 months and 6 months
  Assessed retrospectively (last 1 month) with self-designed question

OTHER OUTCOMES:
Qualitative interviews | 1 month and 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Charite University, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Figura HM, Saha FJ, Seibt S, Haller H, Bringmann HC, Kessler CS, Kugler J, Cramer H, Michalsen A, Kandil FI, Jeitler M. Effects of an Online Meditation Course on Quality of Life and Positive Emotions: A Prospective Observational Study (EXPANSION Study). J Integr Complement Med. 2024 Jun;30(6):518-531. doi: 10.1089/jicm.2023.0099. Epub 2023 Nov 21. PMID 38011030